CLINICAL TRIAL: NCT00352495
Title: A Phase I Study of Vinblastine in Combination With Carboplatin for Children With Newly Diagnosed and Recurrent Low-Grade Gliomas
Brief Title: Vinblastine and Carboplatin in Treating Young Patients With Newly Diagnosed or Recurrent Low-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0515; COG-ADVL0515; CDR0000483184
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors; Neurofibromatosis Type 1
Keywords: childhood low-grade cerebral astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood oligodendroglioma; neurofibromatosis type 1; recurrent childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway and hypothalamic glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neurofibromatosis 1; Astrocytoma; Oligodendroglioma; Optic Nerve Glioma | interventions — Carboplatin; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinblastine sulfate and carboplatin (Experimental): The MTD of vinblastine in combination with a monthly dose of carboplatin will be determined during the first cycle of therapy. Each 4-week cycle will consist of carboplatin once every 4 weeks on day 1. Vinblastine will be given once a week for 3 weeks followed by a one week break. Doses of carboplatin and vinblastine sulfate will be assigned at study enrollment. Patients may receive eleven additional four week cycles, barring tumor progression or unacceptable toxicity. The total duration of therapy will be approximately 48 weeks.
  Interventions: Drug: carboplatin; Drug: vinblastine sulfate

INTERVENTIONS:
Drug: carboplatin
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinblastine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vinblastine when given together with carboplatin in treating young patients with newly diagnosed or recurrent low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the maximum tolerated dose and recommended phase II dose of vinblastine when given in combination with carboplatin in pediatric patients with newly diagnosed or recurrent low-grade gliomas.
* Define and describe the acute and dose-limiting toxicities of this regimen.
* Describe the toxicities associated with repeated courses of the combination chemotherapy regimen and the number of treatment modifications required over the course of treatment.

Secondary

* Describe the radiographic responses in patients treated with this regimen.
* Describe changes in diffusion/perfusion imaging during study therapy.

OUTLINE: This is a multicenter, dose-escalation study of vinblastine. Patients are stratified according to amount of prior therapy (heavily pretreated vs less heavily pretreated).

Patients receive carboplatin IV over 30 minutes on day 1 and vinblastine IV on days 1, 8, 15. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of vinblastine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* low-grade glioma, including 1 of the following subtypes:

  * Astrocytoma variants

    * Fibrillary, protoplasmic, or mixed
  * Pilocytic astrocytoma, including pilomyxoid variants
  * Pleomorphic xanthoastrocytoma
  * Infantile desmoplastic astrocytoma
  * Ganglioglioma
  * Oligodendroglial tumors
  * Mixed glioma, including oligoastrocytoma NOTE: *Biopsy not required for patients who have visual pathway tumors involving the optic nerves and/or optic radiations (i.e., not isolated to the hypothalamus/chiasm)
* Biopsy proven focal low-grade gliomas of the brainstem with measurable disease allowed

  * No diffuse, intrinsic brainstem tumors
* Residual tumor visible on MRI
* Patients without NF-1 must meet the following criteria:

  * Progressive disease after surgery/biopsy based on clear radiographic or clinical evidence of progression OR gross residual tumor (> 1.5 cm²) after surgery/biopsy that is felt to be a high risk to the patient for neurologic and/or visual impairment if the tumor progresses
  * Visual pathway tumors that are not isolated to the hypothalamus/chiasm and are not biopsied must be a high risk to the patient for neurologic and/or visual impairment
* Patients with NF-1 must have evidence of radiographic progression on MRI and/or clinical worsening (e.g., worsening of ophthalmologic exam for visual pathway tumors)
* Meets 1 of the following criteria:

  * Newly diagnosed disease
  * Recurrent disease
* No ventriculoperitoneal shunt-related ascites

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 10 years of age) OR Lansky PS 50-100% (for patients ≤ 10 years of age)
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine based on age, as follows:

  * No greater than 0.8 mg/dL (for patients ≤ 5 years of age)
  * No greater than 1.0 mg/dL (for patients 6-10 years of age)
  * No greater than 1.2 mg/dL (for patients 11-15 years of age)
  * No greater than 1.5 mg/dL (for patients > 15 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal
* ALT ≤ 110 U/L
* Albumin ≥ 2 g/dL
* No history of allergy to carboplatin
* No hyponatremia requiring treatment
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy except for corticosteroids and surgery (for patients with newly diagnosed disease)
* Prior chemotherapy and/or radiotherapy in addition to surgery and corticosteroids allowed (for patients with recurrent disease)
* Prior carboplatin and/or vinblastine allowed if there was no evidence of progressive disease while on therapy and there were no dose reductions due to toxicity (for patients with recurrent disease)
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered (for patients with recurrent disease)
* At least 7 days since prior hematopoietic growth factors (for patients with recurrent disease)
* At least 7 days since prior biological agents (for patients with recurrent disease)
* At least 9 months since prior external beam radiotherapy or gamma knife therapy that included all target lesions (i.e., there is no restriction if a new lesion arises outside the radiation field or a nonirradiated lesion progresses) and recovered (for patients with recurrent disease)
* No other concurrent investigational drugs
* No other concurrent anticancer agents
* No other concurrent chemotherapy, radiotherapy, immunotherapy, or biological therapy
* No concurrent corticosteroids for antiemesis
* Concurrent steroids allowed for tumor edema/increased intracranial pressure provided dose of dexamethasone is stable or decreasing for the past 7 days
* Concurrent physiologic or stress doses of steroids allowed for endocrine deficiencies

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of vinblastine in combination with carboplatin | length of study
Acute and dose-limiting toxicities | length of study
Other toxicities | length of study

SECONDARY OUTCOMES:
Radiographic response | length of study
Changes in diffusion/perfusion imaging | length of study

CONTACTS AND LOCATIONS:
Overall Officials: Regina Jakacki, MD, Study Chair — University of Pittsburgh; Eric Bouffet, MD, MRCP, Study Chair — The Hospital for Sick Children
Locations (21):
- United States (19):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Jakacki RI, Bouffet E, Adamson PC, Pollack IF, Ingle AM, Voss SD, Blaney SM. A phase 1 study of vinblastine in combination with carboplatin for children with low-grade gliomas: a Children's Oncology Group phase 1 consortium study. Neuro Oncol. 2011 Aug;13(8):910-5. doi: 10.1093/neuonc/nor090. Epub 2011 Jul 15. PMID 21764821